CLINICAL TRIAL: NCT05556044
Title: In-hospital Initiation of Empagliflozin for the Treatment of New-onset Acute Heart Failure Regardless of Ejection Fraction: A Pilot Study
Brief Title: Empagliflozin for New On-set Heart Failure Study Regardless of Ejection Fraction
Acronym: EMPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Bryan Ping Yen YAN, Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021.717-T
Record Dates: First submitted 2022-09-15; First posted 2022-09-27 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-02

CONDITIONS: Acute Heart Failure
MeSH Terms: interventions — empagliflozin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Empagliflozin 10 MG (Other)
  Interventions: Drug: Empagliflozin 10 MG

INTERVENTIONS:
Drug: Empagliflozin 10 MG — This is an investigator-initiated, prospective, single-centre, non-randomized open label study that evaluates the efficacy and safety of initiating empagliflozin during index hospitalization for acute heart failure regardless of LVEF.

SUMMARY:
Heart failure (HF) is one of the most important reasons for hospital admission and is associated with high mortality and morbidity. After discharge, up to 40% of patients are readmitted within 6 months and 1-year post-discharge mortality is high. The cost burden of treating patients with HF is high and ~80% of healthcare costs are related to hospital admissions.

Sodium-glucose cotransporter-2 (SGLT2) inhibitor is considered one of the four foundational therapies (ACE-I or ARNI, beta-blockers, MRA, and SGLT2 inhibitors) for HFrEF. In particular, empagliflozin has been shown in randomized controlled trials to reduce the combined risk of cardiovascular death or HF hospitalization in HF patients with both reduced ejection fraction (HFrEF) and preserved ejection fraction (HFpEF). However, guidelines do not specify the sequence and the timing of which therapy to be commenced. The timing of SGLT inhibitors initiation in the treatment of acute HF is not established. In particular, new-onset acute HF is a group which is understudied in the major trials to date. This study aims to evaluate the efficacy and safety of in-hospital initiation of empagliflozin in patients hospitalized for new onset acute HF, regardless of LVEF for up to 90 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Subject age >18 hospitalized for primary diagnosis of acute HF
* Dyspnoea (exertional or at rest) and 2 of the following signs: Congestion on chest X-ray; Rales on chest auscultation; Clinically relevant oedema (e.g. ≥1+ on a 0 to 3+ scale); Elevated jugular venous pressure
* Stabilization criteria (while in the hospital): systolic blood pressure ≥100mmHg and no symptoms of hypotension in the preceding 24 hours; No increase in i.v. diuretic dose for 24 h prior; No i.v. vasodilators including nitrates within the last 24 h prior; No i.v. inotropic drugs for 24 h prior
* NT-proBNP ≥1600 pg/mL or BNP ≥400 pg/mL. (Patients with atrial fibrillation: NT-proBNP ≥2400 pg/mL or BNP

  ≥600 pg/mL. Measured during index hospitalization
* Heart failure hospitalization that requires the treatment of a minimum single dose of 40 mg of i.v.

furosemide( or Equivalent i.v loop diuretics defined as 20 mg of torsemide or 1mg of bumetanide)

Exclusion Criteria:

* Cardiogenic shock
* Documented history of HF with previous HF admission
* Current hospitalization for acute HF primarily triggered by pulmonary embolism, cerebrovascular accident, or acute myocardial infraction
* Interventions in the past 30 days prior or planned during the study: Major cardiac surgery, or Transcatheter aortic valve implantation (TAVI), or percutaneous coronary intervention (PCI), or MitraClip; Implantation of cardiac resynchronization therapy device; Cardiac mechanical support implantation
* Current or expected heart transplant, left ventricular assist device (LVAD), intraaortic balloon pumping (IABP), or patients with planned inotropic support in an outpatient setting
* Haemodynamically severe uncorrected primary cardiac valvular disease planned for surgery or intervention during the course of the study
* eGFR <20 mL/min/1.73m2 as measured during index hospitalization (latest measurement before randomization) or patients requiring dialysis
* Type 1 diabetes mellitus (DM)
* History of ketoacidosis, including diabetic ketoacidosis
* Current or prior treatment with SGLT2 inhibitors in the 90 days prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Heart failure (HF) events | 90 days
  Number of heart failure events (including hospitalization for HFs, urgent heart failure visits and unplanned outpatient visits), time to first heart failure event.
All-cause mortality | 90 days
  All-cause mortality after 90 days of treatment

SECONDARY OUTCOMES:
Change in Kansas City Cardiomyopathy Questionnaire - Total Symptom Score (KCCQ-TSS) | 90 days
  Change from baseline in KCCQ-TSS. Scores are transformed to a range of 0-100, where higher scores reflect better health status.
NT-proBNP level | 90 days
  Change from baseline in log-transformed NT-proBNP level
New York Heart Association (NYHA) class | 90 days
  Change in NYHA class (I-IV), Class IV is most severe; Class I least severe
Major Adverse Cardiovascular Event (MACE) | 90 days
  Measure the occurrence of MACE, including Days alive and out of hospital, occurrence of hypertensive Heart failure from study drug initiation until 90 days after initial hospital discharge and randomization; Time to first occurrence of cardiovascular death or heart failure event until end of trial visit
Occurrence of kidney damage | 90 days
  Occurrence of chronic dialysis or renal transplant or sustained reduction of ≥40% estimated glomerular filtration rate (eGFR), or
  * Sustained eGFR <15mL/min/1.73m2 for patients with baseline eGFR ≥30 mL/min/1.73m2
  * Sustained eGFR <10mL/min/1.73m2 for patients with baseline eGFR <30 mL/min/1.73m2.
Weight loss | 90 days
  Weight loss per mean daily loop diuretic dose after 15, 30, 60 and 90 days of treatment.
Quality-adjusted life years (QALY) gained | 90 days
  Quality-adjusted life years (QALY) gained due to early initiation of empagliflozin
Change in 6 minute hall walk (6MHW) | 90 days
  Change from baseline in 6MHW result

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Yan, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Shatin, Hong Kong

DOCUMENTS (1):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT05556044/Prot_000.pdf